CLINICAL TRIAL: NCT03536871
Title: Exercise and Nutritional Supplementation for Aging and Sedentary Lifestyles
Brief Title: Exercise and Nutritional Supplementation
Acronym: ENSASL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mark Tarnopolsky, Principal Investigator, Professor, Director of Neuromuscular and Neurometabolic Clinic, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4656
Record Dates: First submitted 2018-05-10; First posted 2018-05-25 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia; Healthy Elderly; Healthy Young
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The nutritional supplement will be delivered to a 3rd party contract research organization and the allocation will only be un-blinded after data lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multinutrient Supplement (Active Comparator): Participants will be allocated in a randomized double-masked manner to receive a multi-nutrient supplement (protein and creatine sachet and omega-3 oil) or placebo during a 12 week home-based exercise program and we will assess the influence on the primary and secondary outcomes.
  Interventions: Dietary Supplement: multi-nutrient supplement
- Age biological and chronological (No Intervention): The primary and secondary outcomes will be compared between the younger and older age groups as a function of both exercise and nutritional supplementation.
- Sarcopenia grades (No Intervention): The baseline primary and secondary outcomes will be compared for each of the 3 older adults males groups as a function of muscle mass (healthy active, mild sarcopenia and moderate sarcopenia).
- Exercise - home based programme (Experimental): Each of the older participants will undergo a 12 week home-based exercise program (endurance = increased steps; resistance = body weight and elastic band exercise) to determine the effects on the primary and secondary outcomes.
  Interventions: Other: Exercise

INTERVENTIONS:
Dietary Supplement: multi-nutrient supplement — Compare the effects of a multi-nutrient supplement following a healthy lifestyles program in healthy young men and women, healthy older men, and sarcopenic older men.
  Arms: Multinutrient Supplement
Other: Exercise — We will evaluate the effect of 12 weeks of combined endurance and resistance home-based exercise in younger and older adults.
  Arms: Exercise - home based programme

SUMMARY:
To understand the effects of a novel dietary supplement when used in conjunction with a healthy lifestyle exercise program and to define biomarkers that are specific to sarcopenia. A primary aim in the present study is to determine whether a relationship exists between positive changes in body composition through increases in lean mass and reductions in body fat following oral supplementation of naturally occurring food components in combination with exercise. The purpose of the present study is to examine the effects of a multi-nutrient supplement in combination with an endurance and resistance based exercise intervention in a cohort of older adult men with varying degrees of sarcopenia as compared to younger male controls (McMaster/CIHR/Exerkine project). A sub-purpose nested within the study is to provide serum and muscle samples for use in an aging/sarcopenia biomarker discovery study taken at pre-intervention for the young and older men (Buck Institute/Astellas project).

DETAILED DESCRIPTION:
The present study is a randomized double-blind placebo controlled repeated measures design, with sampling of the cohorts on multiple occasions. Upon obtaining informed consent participants will be randomized into one of six groups:

Healthy younger males - n=20; Healthy older males - placebo n=10, supplement n=10; Sarcopenic older males, placebo, n=20, supplement n=20;

Take home resistance training program The older adult male groups will be provided with a progressive resistance training program which will use exercise bands (Therabands®, Akron, Ohio) and consist of six upper body and six lower body exercises, which will be performed three times per week for 12 weeks without supervision at home. Each session will consist of active warm-up (5min), resistance training with elastic tubing (45min), and cool down (5min). Briefly, the resistance exercises will be performed using elastic tubing for chair squats, hip flexions, leg extensions, leg flexions, ankle dorsiflexion, wall push-ups, back rows, shoulder abductions, triceps extensions, and forearm flexions. Ankle plantar-flexions and abdominal curl-ups will be performed using body weight as resistance. Each participant will be given an exercise instruction booklet and a set of five elastic tubes offering different resistances. Prior to beginning the program trained staff will meet with participants and will teach them how to properly perform exercises in addition to determining the starting elastic tubing size. Furthermore, participants will perform one set of each exercise during weeks 1 and 2, two sets of each exercise during weeks 3 and 4, and three sets of lower body and two sets of upper body exercises during the remaining weeks. Participants will be instructed to move to the next larger tubing size when they can perform 12 repetitions with good exercise form during their last set. This progression will be monitored by the project staff mid way through the study over the phone.

Study products Study products will be provided by Infinit Nutrition Canada (Windsor, Ontario) to all older male subjects, however the young males will only act as baseline controls. The composition of the study products is displayed above in the general experimental design. Both products are similar in taste and appearance and provide an energetic value of ∼200 kcal per serving in a volume of 200 mL. Participants will be asked to consume 1 serving daily of the study product throughout the 12-wk intervention period. Participants will consume their serving at approximately the same time of day, but preferably before breakfast. Participants will be instructed to consume the supplement as a single bolus within 5-10 min. Subjects will also also be provided an omega-3 supplement (or placebo, if they are assigned to the placebo arm) and be instructed to consume 2 teaspoons at the same time as their nutritional supplement. Participants will be instructed to record product intake in a diary to check compliance. To maintain the double-blind nature of the experiment, the placebos, which contains microcrystalline cellulose or safflower oil, will be matched in size and appearance.

Three day weighed food record Participants will be asked to record everything that they consumed for 3 nonconsecutive days: 2 week-days and either a Saturday or a Sunday. On completion of the food record, it will be analyzed using a commercially available computerized database software (Nutribase version 11.5, Cybersoft Inc., Phoenix, AZ, USA). Food items will be aggregated into the following categories: fruit (e.g., fresh/frozen, tinned, juice), vegetables (e.g., fresh/frozen, canned), dairy products (e.g., milk, yoghurt, cheese), breads and cereals (e.g., bread, breakfast cereal, rice, pasta), meats and alternatives (e.g., red meat, poultry, fish, pork, processed meat, tofu, eggs, nuts) and extra foods (e.g., hamburger, pizza, meat pies, chocolate, cake, ice cream, jam, biscuits, crackers, crisps, alcohol).

Pedometer Participants will be given a wearable activity tracker, and instructed on weight training days to aim for 5,000 steps and on all other days to try and reach 10,000. All participants will record their daily totals for subsequent analysis.

Dual X-ray absorptiometry (DXA) and blood pressure A DXA scan is a non-invasive procedure requiring the participant to only lay still on a padded table. It is a fast procedure that provides a variety of body composition variables (bone mass/area/density, fat mass, and fat free mass). The DXA scan exposes individuals to low levels of radiation, approximately 0.18 millirem. According to the United States Nuclear Regulatory Commission, Americans receive approximately 620 millirem each year, half of which is due to environmental background radiation. Radiation exposure can be due to medical treatments or procedures, like X-Ray or MRI's, food, sun exposure, etc. Any exposure to radiation can increase the risk of cancer. In the present study, body composition will be assessed using DXA scan (GE Lunar Prodigy, Madison, WI) and a software program for adults (encore Version 9.15.010). Fat free mass (FFM), fat mass (FM) and bone mineral density (BMD) of the entire body will be recorded. Arterial blood pressure (i.e., systolic [SBP] and diastolic [DBP]) will be measured during rest with a stethoscope (Marshall Nurse Stethoscope, Riverside, Ill., USA) and sphygmomanometer (MDF Instruments Direct Inc., Agoura Hills, Calif., USA).

Muscle biopsies Participants will arrive in the morning in the fasted state and rest quietly in the supine position for 10 minutes. A muscle biopsy will then be taken from the vastus lateralis using local anaesthetic. Samples will be dissected free of connective tissue and immediately partitioned for subsequent analysis (~ 25 mg) for RNA, a small piece (~ 10 mg) will be placed into chilled glutaraldehyde for subsequent electron microscopic evaluation, ~ 20 mg will be frozen for mtDNA deletions, and ~ 50 mg will be frozen for enzyme and protein analysis. The investigators will measure muscle anabolic signaling as previously reported.

Blood sampling A total of 100 mL blood will be taken from the antecubital vein and drawn into evacuated tubes with heparin used for plasma collection and non-treated tubes will be used to collect serum.

Waist and hip circumference measures For waist circumference measurement, the participant will stand with arms at the sides, feet together, and abdomen relaxed. Using a Gulick tape measure, a horizontal measure will be taken at the narrowest part of the torso (above the umbilicus and below the xiphoid process). Obtaining a horizontal measure directly above the iliac crest enhances standardization according to The National Obesity Task Force. For hip circumference measurement, the participant stands erect and feet together, a horizontal measure is taken at the maximal circumference of buttocks.

Physical performance battery A total of four functional tasks will be performed once using a stopwatch that records times to an accuracy 1/100 of a second. First, the 6-minute walk test will involve participants walking as fast as possible around a 20m track for 6 minutes and distance will be measured to the closest meter. Next, the standard 4-stair climb test will involve participants climbing 4 stairs as fast as possible. A 5x sit-to-stand test will involve participants performing a series of consecutive rising and sitting positions from a sturdy, armless plastic chair secured against a wall and with arms crossed at the chest. Finally, the chair rise-and-walk test will involve participants starting from a seated position, standing up and walking as quickly as possible in a predetermined straight line to a pylon 9.14m, while going around the pylon, and returning to their original seated position.

Leg press 1RM Assessment procedures for determining lower body strength using leg press exercise equipment (Cybex Eagle ®, Medway, MA) will require the participant to sit in the leg press machine with the right foot and left foot on the weight platform. The seat and back pad will be adjusted so that feet are flat on the platform hip-width apart, toes slightly angled out, and legs parallel to each other. The interviewer will then instruct the participant to grasp the handles or sides of the seat and extend their legs leaving just a slight bend in the knee. Next, the participant will remove the racking mechanism from the platform and grasp the handles or seat again. The participant will begin with a selected weight that is within their perceived ability, approximately 60 to 80% of maximum capacity (make an educated guess). The participant will lower the platform slowly and controlled towards the chest, keeping the hips and buttocks on the seat, and the back flat against the back pad. Once the thighs are parallel to the platform the participant will extend the legs, pushing the weight back to the start position as hard and as fast as possible. The participant will be instructed to not allow their hips to shift to one side, the buttocks to rise, or knees to move inward or outward during this exercise. The interviewer will also instruct the participant to keep heels flat and not allow the knees to go beyond the toes. Once the repetitions are completed, the participant will replace the racking mechanism and exit the leg press. These procedures were adapted from procedures described by the National Strength and Condition Association (2008) and the American College of Sports Medicine (2013).

Hand grip strength (MVIC) Hand grip strength will be measured using an isometric dynamometer (JAMAR®, Sammons, Bolingbrook, IL). The grip width will be adjusted to hand size and with arm flexed at 90°, the participant will perform three X 5 s efforts with a one min rest between trials.

Knee extension (MVIC) Isometric knee extension will be measured by mechanical dynamometry (Biodex System 3, Biodex Medical Systems, Shirley, NY). Participants will be positioned into the machine with the knee flexed at 90° and perform three X 5s maximal voluntary contractions with 30s rest between each trial.

SF-36 Quality of health Questionnaire The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.

ELIGIBILITY:
Inclusion Criteria:

* Inactive younger men (< 1 hour of formal exercise/week) in the overweight BMI category (25 - 29.9 kg/m2).
* Healthy older male participants will have a body mass index < 30 kg/m2, muscle mass index > 7.23 kg/m2, and a 4-meter walk test > 0.8 m/s.
* Men in the older adult "sarcopenia" group will be individuals that have a body mass index < 30 kg/m2, a muscle mass index between 8.51-10.75 kg/m2, and a 4-meter walk test < 0.8m/s.

Exclusion Criteria:

* Current smokers
* On more than one anti-diabetic drug
* Cardiovascular disease (myocardial infarction and/or hypertension requiring more than 2 medications)
* Congestive heart failure
* Renal disease (creatinine > 130)
* Previous stroke
* Hypertension requiring more than two-pharmacological agents
* Active musculoskeletal injuries and/or severe osteoarthritis
* Significant weight loss in the 3-month period prior to the study
* Vegan diet
* Dairy protein allergy
* History of muscle and/or bone wasting diseases
* Concurrent medications known to affect protein metabolism (i.e. corticosteroids, or prescription strength acne medications)
* Inability to consent
* Chronic obstructive pulmonary disease (FVC or FEV1 < 80% of age predicted mean value or requiring any medication other than a puffer as needed)
* Concurrent supplementation with a dietary protein, calcium, l-leucine, creatine, CoQ10, alpha lipoic acid, n-3 PUFA, and conjugated linoleic acid.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Body Composition | 12 weeks
  Fat-Free and Fat Mass
Muscle Strength | 12 weeks
  Knee extension isometric strength and leg press
Functional Outcomes | 12 weeks
  6 Minute Walk Test

SECONDARY OUTCOMES:
Mitochondrial Function | 12 weeks
  COX IV Enzyme Activity
Muscle Fibre Size | 12 weeks
  Type I and II fibre size
Inflammatory markers | 12 weeks
  IL-6
Quality of Life assessment | 12 weeks
  SF-36 questionnaire
Glycemia measurements | 12 weeks
  hemoglobin A1C
Plasma lipids | 12 weeks
  Cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Mark Tarnopololsky, MD/PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brose A, Parise G, Tarnopolsky MA. Creatine supplementation enhances isometric strength and body composition improvements following strength exercise training in older adults. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):11-9. doi: 10.1093/gerona/58.1.b11. PMID 12560406
- [Result] Tarnopolsky M, Zimmer A, Paikin J, Safdar A, Aboud A, Pearce E, Roy B, Doherty T. Creatine monohydrate and conjugated linoleic acid improve strength and body composition following resistance exercise in older adults. PLoS One. 2007 Oct 3;2(10):e991. doi: 10.1371/journal.pone.0000991. PMID 17912368
- [Result] Bell KE, Snijders T, Zulyniak M, Kumbhare D, Parise G, Chabowski A, Phillips SM. A whey protein-based multi-ingredient nutritional supplement stimulates gains in lean body mass and strength in healthy older men: A randomized controlled trial. PLoS One. 2017 Jul 18;12(7):e0181387. doi: 10.1371/journal.pone.0181387. eCollection 2017. PMID 28719669
- [Result] Murphy CH, Saddler NI, Devries MC, McGlory C, Baker SK, Phillips SM. Leucine supplementation enhances integrative myofibrillar protein synthesis in free-living older men consuming lower- and higher-protein diets: a parallel-group crossover study. Am J Clin Nutr. 2016 Dec;104(6):1594-1606. doi: 10.3945/ajcn.116.136424. Epub 2016 Nov 9. PMID 27935521
- [Result] Churchward-Venne TA, Breen L, Di Donato DM, Hector AJ, Mitchell CJ, Moore DR, Stellingwerff T, Breuille D, Offord EA, Baker SK, Phillips SM. Leucine supplementation of a low-protein mixed macronutrient beverage enhances myofibrillar protein synthesis in young men: a double-blind, randomized trial. Am J Clin Nutr. 2014 Feb;99(2):276-86. doi: 10.3945/ajcn.113.068775. Epub 2013 Nov 27. PMID 24284442
- [Result] Nilsson MI, Mikhail A, Lan L, Di Carlo A, Hamilton B, Barnard K, Hettinga BP, Hatcher E, Tarnopolsky MG, Nederveen JP, Bujak AL, May L, Tarnopolsky MA. A Five-Ingredient Nutritional Supplement and Home-Based Resistance Exercise Improve Lean Mass and Strength in Free-Living Elderly. Nutrients. 2020 Aug 10;12(8):2391. doi: 10.3390/nu12082391. PMID 32785021
- [Result] Perez K, Ciotlos S, McGirr J, Limbad C, Doi R, Nederveen JP, Nilsson MI, Winer DA, Evans W, Tarnopolsky M, Campisi J, Melov S. Single nuclei profiling identifies cell specific markers of skeletal muscle aging, frailty, and senescence. Aging (Albany NY). 2022 Dec 13;14(23):9393-9422. doi: 10.18632/aging.204435. Epub 2022 Dec 13. PMID 36516485
- See also: Pubmed link primary publication (Nilsson et al.) — http://pubmed.ncbi.nlm.nih.gov/32785021/
- See also: Pubmed link to aging biomarker publication (Perez et al.) — https://pubmed.ncbi.nlm.nih.gov/36516485/